CLINICAL TRIAL: NCT02779439
Title: Therapeutic Infusion of Partially HLA-matched Third Party Donor-derived Virus- and Fungus Specific T-lymphocytes in Patients With Active Viral or Fungal Infection Post-allogeneic Stem Cell or Solid Organ Transplantation
Brief Title: Partially HLA-matched Third Party Antigen Specific T-cells for Infection Post-stem Cell or Solid Organ Transplantation
Acronym: R3ACT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sydney (Other)
Responsible Party: Principal Investigator, David Gottlieb, Professor David Gottlieb, University of Sydney
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R3ACT
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: CMV Infection; EBV; Adenovirus
MeSH Terms: conditions — Cytomegalovirus Infections; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3rd party CTL infusion (Experimental): Virus specific CTLs
  Interventions: Biological: Virus specific CTLs

INTERVENTIONS:
Biological: Virus specific CTLs — Virus specific CTLs will be given to patients with persistent or recurrent viral reactivation after 2 weeks of standard anti-viral therapy
  Other Names: T cells

SUMMARY:
To assess the safety and biological efficacy of therapeutically administered most closely HLA-matched third party donor-derived specific cytotoxic T lymphocytes (CTLs) targeting cytomegalovirus (CMV) or Adenovirus (Adv) or Epstein Barr virus (EBV) or fungi including Aspergillus and Candida species for the treatment of viral infection following allogeneic blood or marrow stem cell or solid organ transplantation.

DETAILED DESCRIPTION:
The study will analyse the safety and biological efficacy of administering the investigational products (most closely HLA-matched third party donor-derived T cells stimulated with viral or fungal antigen expressing DC), for the treatment of viral reactivation and/or infection or fungal infection following allogeneic blood or marrow or solid organ transplantation. The cells will be given therapeutically after transplantation in patients with active viral reactivation or proven/probably fungal infection despite standard therapy.

Our AIMS are to study the safety of third party donor-derived CTL infusions, their effect on treatment of viral reactivation as well as their effect on reconstitution of virus- and fungus-specific immunity, viral and fungal infection and reactivation rates after transplantation, viral load, and use of antiviral and antifungal pharmacotherapy.

We will evaluate the safety of infusions with respect to the development of adverse events within the first 12 months post-CTL infusion and the dynamics of cell persistence by T-cell chimerism analysis.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of myeloablative or non-myeloablative allogeneic or solid organ transplantation for any indication.
* Presence of viral reactivation or infection with CMV, Adv or EBV or invasive fungal disease must be present at the time of infusion as determined by:

  * For CMV CMV detectable by antigen detection, PCR or culture in peripheral blood or tissue biopsy or by immunohistochemical staining on tissue biopsy specimen
  * For Adv Presence of Adv as detected by PCR, antigen detection or culture in body fluids including blood, stool, urine or nasopharyngeal secretions
  * For EBV Elevated EB virus detectable in peripheral blood by PCR or Presence of documented EBV related PTLD diagnosed by tissue biopsy or Elevated EB virus detectable in the blood by PCR and clinical or imaging findings consistent with EBV lymphoma
  * For invasive fungal disease Proven or probable invasive fungal disease according to De Pauw 2008[114]
* Failure of standard therapy as defined by:

  * For CMV The continued presence of detectable CMV virus or antigen after at least 14 days of antiviral therapy with IV ganciclovir or foscarnet Recurrence of detectable CMV virus or antigen after at least 2 weeks of prior antiviral therapy
  * For Adv A rise or less than 50% reduction in viral load in blood or any site of disease as measured by PCR or any quantitative assay despite use of therapy as determined by the treating physician; Standard therapy may include intravenous cidofovir within the limits of renal function
  * For EBV Increase or less than 50% decrease in the size of EBV lymphoma or

Increase or less than 50% decrease in the EBV viral load in peripheral blood despite use of appropriate therapy as determined by the treating physician which may include:

* Reduction in immunosuppression
* Rituximab 375mg/m2 up to 4 infusions
* Cytotoxic chemotherapy

  o For invasive fungal disease inadequate or incomplete clinical response according to treating physician after at least 5 days of best available therapy
* Adequate hepatic and renal function (< 3 x upper limit of normal for AST (SGOT), ALT (SGPT), < 2 x upper limit of normal for total bilirubin, serum creatinine)
* ECOG status 0 to 3 or Lansky score 30-100
* Patient (or legal representative) has given informed consent

Exclusion Criteria:

* Use of anti-lymphocyte globulin (ALG, ATG, Campath or other broad spectrum lymphocyte antibody) given in the 4 weeks immediately prior to infusion or planned within 4 weeks after infusion.
* Grade II or greater graft versus host disease within 1 week prior to infusion.
* Prednisone or methylprednisolone at a dose of > 1 mg/kg (or equivalent in other steroid preparations) administered within 72 hours prior to cell infusion.
* ECOG status 4 or Lansky score <30
* Privately insured in or outpatients in New South Wales participating centres (see 12.5 Indemnity issues).

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Infusion related safety | 1 week
  infusion related adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Westmead Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Withers B, Blyth E, Clancy LE, Yong A, Fraser C, Burgess J, Simms R, Brown R, Kliman D, Dubosq MC, Bishop D, Sutrave G, Ma CKK, Shaw PJ, Micklethwaite KP, Gottlieb DJ. Long-term control of recurrent or refractory viral infections after allogeneic HSCT with third-party virus-specific T cells. Blood Adv. 2017 Nov 2;1(24):2193-2205. doi: 10.1182/bloodadvances.2017010223. eCollection 2017 Nov 14. PMID 29296867